CLINICAL TRIAL: NCT03492229
Title: Cortical Priming to Optimize Gait Rehabilitation Post Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sangeetha Madhavan, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011-0676; R01HD075777 (NIH)
Record Dates: First submitted 2018-03-09; First posted 2018-04-10 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Stroke
Keywords: Gait; Brain stimulation; tDCS; Walking
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tDCS+AMT (Experimental): TDCS in combination with movement training before treadmill training
  Interventions: Other: tDCS; Other: AMT; Behavioral: Treadmill training
- tDCS (Active Comparator): tDCS only before treadmill training
  Interventions: Other: tDCS; Behavioral: Treadmill training
- AMT (Active Comparator): Movement training only before treadmill training
  Interventions: Other: AMT; Behavioral: Treadmill training
- Control (Sham Comparator): No priming before treadmill training
  Interventions: Behavioral: Treadmill training

INTERVENTIONS:
Other: tDCS — 1 mA of tDCS
  Arms: tDCS; tDCS+AMT
Other: AMT — Ankle motor training
  Arms: AMT; tDCS+AMT
Behavioral: Treadmill training — High intensity treadmill training

SUMMARY:
Over four million stroke survivors currently living in the United States are unable to walk independently in the community. To increase the effectiveness of gait rehabilitation, it is critical to develop therapies that are based on an understanding of brain adaptations that occur after stroke. This project will be the first step towards the development of a novel therapeutic approach using brain stimulation to increase walking capacity in stroke survivors and understand the neural mechanisms that are associated with impairment and functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 - 80 years
* First ever monohemispheric stroke > 6 months since onset
* Residual hemiparetic gait deficits
* Able to walk without an ankle orthotic for 5 minutes at self-paced speed. Handheld assistive device is acceptable.

Exclusion Criteria:

* Severe osteoporosis
* Contracture-limiting range of motion of lower limb
* Uncontrolled anti-spasticity medications during the study period
* Cardiorespiratory or metabolic diseases (e.g. cardiac arrhythmia, uncontrolled hypertension or diabetes, chronic emphysema)
* Unhealed decubiti, persistent infection
* Significant cognitive or communication impairment (MMSE <21), which could impede the understanding of the purpose of procedures of the study or prevent the patient from performing the tracking task.
* Lesions pertaining to the brainstem and cerebellum

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Change in gait speed using 10 meter walk test | Change from baseline to immediately after training and baseline to 3 months follow up
  10-meter walk test: Gait speed will be measured as the average of 3 trials of the 10-m walk test. Participants will be asked to walk at their normal comfortable pace to cover a distance of 10 meters without an AFO (handheld assistive device is acceptable if needed).

SECONDARY OUTCOMES:
Change in 6 minute walk test | Change from baseline to immediately after training and baseline to 3 months follow up
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. Participants will be asked to walk at their normal pace for 6 minutes.
Change in Berg Balance Scale | Change from baseline to immediately after training and baseline to 3 months follow up
  Balance will be measured using the Berg Balance Scale. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function. Tasks such as standing with eyes closed, one leg stance etc are included.
Change in Quality of life measures | Change from baseline to immediately after training and baseline to 3 months follow up
  QOL will be measured with the Stroke Impact Scale (SIS). The SIS is a stroke-specific self-reported health status measure.
Change in cortical excitability of leg muscles using TMS | Change from baseline to immediately after training and baseline to 3 months follow up
  Transcranial magnetic stimulation will be used to measure contralateral and ipsilateral corticospinal excitability of the paretic tibialis anterior (TA) using the protocol previously published by the PI Dr. Madhavan.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeetha Madhavan, Principal Investigator — UIC
Locations (1):
- The University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madhavan S, Cleland BT, Sivaramakrishnan A, Freels S, Lim H, Testai FD, Corcos DM. Cortical priming strategies for gait training after stroke: a controlled, stratified trial. J Neuroeng Rehabil. 2020 Aug 17;17(1):111. doi: 10.1186/s12984-020-00744-9. PMID 32799922